CLINICAL TRIAL: NCT05804747
Title: A Multicenter, Prospective, Non-interventional Study to Evaluate Effectiveness and Safety of Edoxaban in Patients 80 Years of Age or Older With Nonvalvular Atrial Fibrillation
Brief Title: A Study to Evaluate Effectiveness and Safety of Edoxaban in Patients 80 Years of Age or Older With Nonvalvular Atrial Fibrillation
Acronym: SILVERCARE_AF
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LIX-OS-22-01
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
Keywords: Non-valvular Atrial fibrillation; Elderly Patients
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Edoxaban: Participants who were prescribed edoxaban within 8 weeks of study enrollment at the discretion of the physician and were prospectively followed to assess the efficacy and safety of prescribed edoxaban.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — This is observational, non-interventional study. No study drug will be administered during this study.

SUMMARY:
Non-valvular atrial fibrillation (NVAF) increases the risk of stroke by three- to five-fold, especially in elderly patients, creating a huge burden on medical system as well as a negative impact on patients' lives. Direct oral anticoagulants (DOACs) are recommended for patients with NVAF to prevent strokes. Real world data reveal the underuse of anticoagulation in the elderly, especially due to physicians' concern of bleeding, often neglecting the thromboembolic risk. This study is designed to evaluate the safety and effectiveness of edoxaban in Korean elderly patients with atrial fibrillation.

DETAILED DESCRIPTION:
The objective of this study will be to evaluate the safety and effectiveness of edoxaban in patients 80 years of age or older with NVAF. This observational, non-interventional study will prospectively follow Korean patients who have been prescribed edoxaban at the discretion of the physician up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* NVAF participants aged ≥ 80 years old
* Participants who are determined to be prescribed with edoxaban at the discretion of the physician within 8 weeks prior to enrollment according to Package information
* Participants who can return to the site in person for face-to-face visits
* Written informed consent for participation in the study (ICF)

Exclusion Criteria:

* Planning to participate or simultaneously participating in any interventional study
* Life expectancy < 1 year

No influence on prescribing behavior as participants will only be included in the study after the physicians have made the clinical decision to prescribe edoxaban.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will include participants who are prescribed with edoxaban at the discretion of the physician within 8 weeks prior to enrollment. Data documentation will occur every 6 (± 90 days) and 12 months (± 90 days) from the start of edoxaban treatment. Patient visits will be conducted according to regular clinical care and should not be influenced by the foreseen data documentation time points.
Sampling Method: Non-Probability Sample
Enrollment: 1204 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Composite of Stroke, Systemic Embolic Events, Major Bleeding, or All-Cause Mortality | Baseline up to 12 months

SECONDARY OUTCOMES:
Number of Participants With Composite Events (Stroke, Systemic Embolism, or Cardiovascular Mortality), (Stroke, Systemic Embolism, or All-Cause Mortality), (Stroke [Ischemic, Hemorrhagic] or Systemic Embolism), and (Stroke [Ischemic, Hemorrhagic]) | Baseline up to 12 months
Percentage of Participants With Stroke (Ischemic, Hemorrhagic), Systemic Embolism, Cardiovascular Mortality, and All-Cause Mortality | Baseline up to 12 months
Number of Hospitalizations Related to Cardiovascular Conditions | Baseline up to 12 months
Percentage of Participants With Transient Ischemic Attack, Venous Thromboembolism, and Major Cardiovascular Events | Baseline up to 12 months
Number of Participants With Composite of Stroke, Systemic Embolic Events, Major Bleeding, or All-Cause Mortality, Based on Independent Risk Factors | Baseline up to 12 months
Number of Participants With Bleeding Events (Major, Clinically Relevant Non-Major, Minor, and Composite) | Baseline up to 12 months
Percentage of Participants With Edoxaban Dose Change, Based on Reason for Dose Change | Baseline up to 12 months
Percentage of Participants Who Permanently Discontinued Edoxaban, Based on Reason for Discontinuation | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (33):
- South Korea (33):
  - Korea University Ansan Hospital, Ansan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Samsung Changwon Center, Changwon
  - Dankook University Hospital, Cheonan
  - Soonchunhyang University Hospital, Cheonan
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Catholic University of Korea Daejeon St. Mary's Hospital, Daejeon
  - Chungnam University Hospital, Daejeon
  - National Health Insurance Service Ilsan Hospital, Goyang
  - Chosun University Hospital, Gwangju
  - Chonnam Natinal University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul
  - KyungHee University Hospital at GangDong, Seoul
  - Korea Veterans Health Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hosptial, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Catholic University of Korea St. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No